CLINICAL TRIAL: NCT04173312
Title: Efficacy of Local Anesthetic Through Continuous Infusion Following Laparotomy Procedures.
Brief Title: Efficacy of Local Anesthetic Through Continuous Infusion
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ascension Health (Industry)
Responsible Party: Principal Investigator, Tarik Wasfie, MD, Principle Investigator, Ascension Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AscensionGenesysH
Record Dates: First submitted 2019-11-20; First posted 2019-11-21 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Pain Control
Keywords: local anesthetic; continuous infusion; pain control
MeSH Terms: conditions — Agnosia | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Who Masked: Participant, Investigator
Masking Description: Infusion will be the same for both groups. One will have analgesic and one will have saline.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Infused analgesic (Active Comparator): Patients will be assigned to receive local anesthetic through continuous infusion by pump.
  Interventions: Combination Product: Bupivacaine infusion
- Infused saline (Placebo Comparator): Patients will be assigned to receive saline through continuous infusion by pump.
  Interventions: Combination Product: Saline

INTERVENTIONS:
Combination Product: Bupivacaine infusion — Local systemic Infusion of anesthetic
  Arms: Infused analgesic
Combination Product: Saline — Local systemic infusion of saline
  Arms: Infused saline

SUMMARY:
Efficacy of using continuous infusion of local anesthetic for post operative pain control following laparotomy.

DETAILED DESCRIPTION:
This study will evaluate the benefits of placing an analgesic pain pump in laparotomy incisions with the addition of intravenous/oral pain medications as needed versus using solely intravenous and oral pain medications as needed for post-operative pain management. The goal of this study will be to decrease the usage of narcotics in post-operative laparotomy patients by providing local incision pain relief. This will be a double blinded randomized control study with placebo with two groups of patients: One with a local anesthetic infusion pump filled with Bupivacaine, a local anesthetic, after laparotomy and the other group with an infusion pump filled with normal saline. The pain pumps will be placed in the OR. Post-operatively, all patients will have the standard pain regimen available to them during their stay. Surgeons will monitor the patient for 4 days post-operatively and the infusion pain pump will be removed on post-operative day 4. Investigator will then look back through each patient's records and gather the amount of pain medications that they requested during their stay. Both groups will then have their data collected in the same manner and placed for data analysis. - The standard pain regimen will include a morphine IV 4mg every 4 hours and Hydrocodone-acetominophen 5/325 Q6H PRN. If a patient controlled analgesia infusion pump is needed this will be considered a need for increase in pain management. Every patient will be started on this pain regimen post operatively. During their stay, If the patient requires an increase in their pain medication, the supervising attending will determine which drug will be added in improve their pain. At the end of the patients stay, the amount of narcotic usage will be compiled and turned into morphine equivalents in order to compare them with the control group.

ELIGIBILITY:
Inclusion Criteria:

- Patients scheduled for elective laparotomy

Exclusion Criteria:

* Emergency laparotomy
* Pregnancy
* Patients on chronic pain medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Self Reported Pain | 5 days
  Patient reported pain rating on the Visual Analog Scale (VAS) for Pain. Pain intensity is rated on a scale of 0 to 100. It is anchored by 0 for no pain and 100 for worst pain ever.

CONTACTS AND LOCATIONS:
Overall Officials: Tarik Wasfie, MD, Principal Investigator — Ascension Health
Locations (1):
- Ascension Genesys Hospital, Grand Blanc, Michigan, United States

IPD SHARING:
Plan to Share IPD: No